CLINICAL TRIAL: NCT00416403
Title: Randomized Phase II Biomarker Pilot Trial of Fluvastatin Use in Women With Ductal Carcinoma in Situ (DCIS) or Stage I Breast Cancer
Brief Title: Effect of Fluvastatin on Biomarkers in Women Who Are Undergoing Surgery for Ductal Carcinoma In Situ or Stage I Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDR0000522934; UCSF-047522; UCSF-H8409-26206-01; MSKCC-06041
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: breast cancer in situ; ductal breast carcinoma in situ; stage IA breast cancer; stage IB breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — Fluvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Experimental): Patients receive oral fluvastatin sodium once daily for 3-6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fluvastatin sodium
- Arm II (Experimental): Patients receive oral fluvastatin sodium as in arm I at a higher dose.
  Interventions: Drug: fluvastatin sodium
- Arm III (Experimental): Patients do not receive fluvastatin sodium. breast Cancer surgery only
  Interventions: Procedure: Breast Cancer Surgery Only - Arm III

INTERVENTIONS:
Drug: fluvastatin sodium — Given orally
  Arms: Arm I; Arm II
Procedure: Breast Cancer Surgery Only - Arm III — Breast Cancer Surgery
  Arms: Arm III

SUMMARY:
RATIONALE: Collecting samples of blood and tissue from patients with cancer to study in the laboratory may help doctors learn how fluvastatin effects biomarkers related to breast cancer.

PURPOSE: This randomized phase II trial is studying how fluvastatin effects biomarkers in women undergoing surgery for ductal carcinoma in situ or stage I breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine differences between measures of cell proliferation (Ki-67) in women with ductal carcinoma in situ (DCIS) or stage I breast cancer receiving neoadjuvant fluvastatin sodium.

Secondary

* Determine whether statin use differentially affects specific types of DCIS/early-stage breast cancer (comedo, estrogen receptor [ER]-positive, ER-negative).
* Compare differences between tissue staining of CD68, circulating macrophages, and regulatory T cells in these patients.
* Assess the feasibility of using inherent susceptibility (mRNA polymerase chain reaction testing) to predict response to statins in these patients.

OUTLINE: This is a randomized, controlled, single-blind, multicenter, pilot study. Patients are randomized to 1 of 2 treatment arms (arms I or II). Patients accrued as control participants are assigned to arm III.

* Arm I: Patients receive oral fluvastatin sodium once daily for 3-6 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral fluvastatin sodium as in arm I at a higher dose.
* Arm III (control): Patients do not receive fluvastatin sodium. All patients then undergo definitive surgery.

Patients in arms I and II undergo blood collection at baseline and at the time of surgery for biomarker analysis. Patients in arm III undergo blood collection at baseline and then approximately 1 month later. Tissue is collected from patients in all arms at the time of surgery. Blood and tissue samples are examined for biological markers, including Ki-67, C-reactive protein, cleaved caspase 3, HER2, CD68 gene, and estrogen and progesterone receptors by immunohistochemistry. Markers of inflammation (e.g., comedo necrosis macrophages and CD25-positive T cells), low-density lipoprotein, and cholesterol are also analyzed. Serum mRNA is measured by polymerase chain reaction.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ductal carcinoma in situ (DCIS) or stage I breast cancer by stereotactic core or incisional biopsy
* Planning to undergo surgery in 3-6 weeks

  * Patients undergoing re-excision due to evidence of tumor present at surgical margins are eligible
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* ALT and AST ≤ 10% above upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to tolerate statins
* Willing to undergo 2 blood draws (separated by approximately 3-4 weeks) during study participation (control arm)

PRIOR CONCURRENT THERAPY:

* No other concurrent statins
* No concurrent chemotherapy
* No concurrent administration of any of the following:

  * Niacin
  * Propranolol
  * Cholestyramine
  * Cyclosporine
  * Digoxin
  * Erythromycin
  * Itraconazole
  * Gemfibrozil
  * Phenytoin
  * Diclofenac
  * Tolbutamide
  * Glyburide
  * Losartan
  * Cimetidine
  * Ranitidine
  * Omeprazole
  * Rifampin
  * Warfarin
* No initiation of new hormonal therapy during study participation
* Concurrent participation in other clinical trials (e.g., for DCIS or prevention) is allowed

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-07; Primary Completion 2007-09 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in proliferation after statin exposure, as measured by Ki-67 level | up to 6 weeks

SECONDARY OUTCOMES:
Blood and serum markers, including C-reactive protein, cleaved caspase 3, HER2, CD68, macrophages and immunoregulatory CD25 T cells, estrogen and progesterone receptors, mRNA, low-density lipoprotein, and cholesterol | up to 6 weeks
Presence of comedo necrosis | up to 6 weeks
Safety | up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laura J. Esserman, MD, MBA, Study Chair — University of California, San Francisco
Locations (4):
- United States (4):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Result] Garwood ER, Kumar AS, Baehner FL, Moore DH, Au A, Hylton N, Flowers CI, Garber J, Lesnikoski BA, Hwang ES, Olopade O, Port ER, Campbell M, Esserman LJ. Fluvastatin reduces proliferation and increases apoptosis in women with high grade breast cancer. Breast Cancer Res Treat. 2010 Jan;119(1):137-44. doi: 10.1007/s10549-009-0507-x. PMID 19728082